CLINICAL TRIAL: NCT02198742
Title: A Comparison Between Two Video Laryngoscopes,the Truview PCD and the Glidescope Cobalt AVL, in Successfully Intubating Pediatric Mannequins With and Without Difficult Airways
Brief Title: A Comparison Between Two Video Laryngoscopes,in Successfully Intubating Pediatric Mannequins w/wo Difficult Airways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helena Karlberg, Pediatric Anesthesiologist, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H28224
Record Dates: First submitted 2014-01-15; First posted 2014-07-24 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Miller blade (Active Comparator): Subjects must have >500 intubations in order to participate in this study. There is no placebo group, and each subject wil be his or her own control.
  Interventions: Device: Miller blade
- Truview PCD (Active Comparator): Subjects were given a quick guide of the Truview PCD supplied by the manufacturer with step by step instructions for use. They were also given time to practice with the device on a normal model until they felt comfortable. There is no placebo group, and each subject wil be his or her own control.
  Interventions: Device: Truview PCD
- Glidescope Cobolt (Active Comparator): Subjects were required to watch a instructional video provided by the manufacterer. Subjects were then allowed to practice on a normal model until they felt comfortable before beginning the study. There is no placebo group, and each subject wil be his or her own control.
  Interventions: Device: Glidescope Cobolt

INTERVENTIONS:
Device: Miller blade — To participate in the study the subjects must have >500 intubations with the miller blade.
  Arms: Miller blade
Device: Truview PCD — Subjects were given a quick guide of the Truview PCD supplied by the manufacturer with step by step instructions for use. They were also given time to practice with the device on a normal model until they felt comfortable.
  Other Names: Trueview PCD - Multichoice video laryngoscope system
  Arms: Truview PCD
Device: Glidescope Cobolt — Subjects were required to watch a instructional video provided by the manufacturer. Subjects were then allowed to practice on a normal model until they felt comfortable before beginning the study. There is no placebo group, and each subject wil be his or her own control.
  Arms: Glidescope Cobolt

SUMMARY:
The study is a randomized crossover study where anesthesia practitioners will intubate three different pediatric infant mannequins (normal airway, anterior larynx, Pierre Robin syndrome anatomy) using three different intubation devices (the Miller blade, the Truview VL, the Glidescope Cobalt video-laryngoscope) in two different scenarios (normal neck and with an immobile neck). The order of presentation will be randomized. As this is a cross over study, all subjects will complete all scenarios. There is no placebo group, and each subject wil be his or her own control.

DETAILED DESCRIPTION:
Participants will be given individual, standardized instructions and demonstrations for each device as per the manufacturers' instructions. The participants will practice with instructor's feedback on an infant mannequin with a normal airway until he/she feel comfortable with each of the three devices. The investigator will record the prior experience of the participant in using each of the 3 devices in clinical situations. Each subject will be asked to intubate each of the mannequins with each of the devices. The choice of the order of device and mannequin will be based on a Latin square design and the sequence will be assigned to participants based on a computer generated random number. A closed envelope technique will blind participants and investigators to the order of airway device and mannequin till the start of the individual trial. Participants will first finish the test on unchanged conditions and then repeat the process using the same order of mannequins and devices but with the neck held immobile to simulate a scenario of a child with an unstable cervical spine. Data from different scenarios will be recorded from a total number of 18 attempts of tracheal intubation per participant. Participants will be asked to proceed as though they were in the operating room with an assistant available to follow their commands. The order of presentation of each mannequin, airway device and scenario will be randomized as described above. The time from placing the device in the mannequin's mouth to the time the Ambu bag is connected to the end of the tracheal tube and a positive pressure breath is given will constitute the intubation time. During each intubation the participant will be asked to state when he or she has obtained the best view for intubation and this time this will be recorded as the time for visualization. The subject will assess the quality of the best glottic view on the Cormack - Lehane grade of 1 -4. The investigators will record all maneuvers to optimize visualization of the larynx such as tracheal pressure, lip retraction, pulling the tongue forward etc. The time from entry of the device in the mouth to the time the tracheal tube is started to be advanced is the visualization time. The time a positive pressure breath is given at the end of the tracheal tube will constitute the end of the attempt of intubation. A failed attempt is defined as removal of the laryngoscope from the mouth without a successful intubation. The number of times the endotracheal tube is advanced will also be recorded. Failure of intubation will be defined as unrecognized esophageal intubation, abandoned procedure, intubation taking longer than 120 seconds and intubation requiring more than 3 attempts. The observer will estimate the maximum force applied to the maxilla on a 0 -10 scale where 0= no force and 10 = maximum force with distortion of the maxilla. The observer will also estimate potential damage of laryngeal structures on a 0 -10 scale.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia practitioners including anesthesia attendings, fellows, residents CAIII and CRNA's at Texas Children's Hospital Department of Anesthesiology with clinical experience of >500 intubations with Miller blades.

Exclusion Criteria:

* Anesthesia practitioners with <500 intubations with Miller blades.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time required for successful endotracheal intubation with the three devices. | Subjects complete study in 1 day
  The devices to be compared include (1)the standard Miller blade, (2) the GlideScope Cobalt AVL and (3) the Truview PCD video-laryngoscopes. Successful intubation will be measured in the seconds from the time the recorder says "begin" until time of first positive pressure breath and confirmation endotracheal tube is in the trachea.

SECONDARY OUTCOMES:
Time to visualize the larynx | From time recorder says "begin" till subject rates best view up to 3minutes
  Start time is when the recorder says "begin" . The time to visualize the larynx ends when the subject rates best view of the larynx.
Time from visualization of larynx to tracheal intubation | one day
  time from the beginning of the endotracheal tube being inserted till first positive pressure breath measured in seconds.
Number of attempts at tracheal intubation | one day
  Subjects were allowed a total of 3 attempts at tracheal intubation with a device on a mannequin.
Number of failed attempts | one day
  Subjects were allowed 3 unsuccessful attempts with each device. After 3 unsuccessful attempts with a device the subject was considered to have failed that device.
Amount of force on the maxilla | one day
  Observer rated the amount of force on the maxilla based on a 0-10 point scale. The observer was the same for all cases.
Optimization measures for laryngeal visualization and tracheal intubation | one day
  The subjects were allowed to ask for assistance with optimization such as external tracheal pressure, lip retraction, or pulling on the tongue. All subjects were instructed that no measures would be taken unless asked for and intructed on what assistance was needed. The observer recorded and counted all optimizing measures.
Documentation of participant's comments on preference of device | one day
  All participants were asked at the completion of the study what device they prefered for a case with anticipated difficult intubation. A count was made of their preference.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Karlberg, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children't Hospital, Houston, Texas, United States